CLINICAL TRIAL: NCT02972502
Title: Investigating the Efficacy of Using Haloperidol vs. Metoclopramide for Treatment of Acute Headaches and Migraines in the Emergency Department: A Prospective Randomized Clinical Trial
Brief Title: Efficacy of Haloperidol vs. Metoclopramide for Treatment of Acute Headaches and Migraines in the Emergency Department
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: PI lapsed institutional training
Sponsor: OhioHealth (Other)
Responsible Party: Principal Investigator, Christopher Lloyd, Attending Physician, OhioHealth
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-0078
Record Dates: First submitted 2016-11-07; First posted 2016-11-23 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-09

CONDITIONS: Headache, Migraine
Keywords: Metoclopramide (Reglan); Haloperidol (Haldol)
MeSH Terms: conditions — Migraine Disorders | interventions — Metoclopramide; Haloperidol; Saline Solution; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metoclopramide (Reglan) (Active Comparator): Patients will receive 10 mg of intravenous (IV) metoclopramide following a 1-liter bolus of normal saline (NS) and 25 mg of IV diphenhydramine.
  Interventions: Drug: Metoclopramide; Other: Normal Saline; Drug: Diphenhydramine
- Haloperidol (Haldol) (Experimental): Patients will receive 2.5 mg of intravenous (IV) haloperidol following a 1-liter bolus of normal saline (NS) and 25 mg of IV diphenhydramine.
  Interventions: Drug: Haloperidol; Other: Normal Saline; Drug: Diphenhydramine

INTERVENTIONS:
Drug: Metoclopramide — Patients receive 10 mg of intravenous (IV) metoclopramide.
  Other Names: Reglan
  Arms: Metoclopramide (Reglan)
Drug: Haloperidol — Patients receive 2.5 mg of IV haloperidol.
  Other Names: Haldol
  Arms: Haloperidol (Haldol)
Other: Normal Saline — All patients receive a 1-liter bolus of normal saline (NS)
Drug: Diphenhydramine — All patients receive 25 mg of intravenous (IV) diphenhydramine.
  Other Names: Benadryl

SUMMARY:
Metoclopramide (Reglan) is a common agent used for relief of headaches in the emergency department (ED).In this study the investigators seek to explore another option for treatment of headaches in the ED, one that may be more efficacious and efficient. Haloperidol (Haldol), a butyrophenone class of medication, is thought to act by affecting the dopamine 2 receptor in the brain.

By exploring haloperidol as an option for treatment, the investigators hope to discover a more efficient and effective medication for the treatment of non-traumatic headaches, thereby decreasing a patient's length of stay in the department and decreasing the rate of return visits for continued discomfort from the same headache. This study could lead to the increased usage of haloperidol as a first line agent in the treatment of prolonged headaches presenting to the ED.

DETAILED DESCRIPTION:
At this time, choice of medications for the treatment of headaches in the ED is still based on personal and patient preferences because no properly constructed trials have been carried out that would allow identification of a superior agent. Metoclopramide (Reglan) is a common agent used for relief of headaches in the ED. Uncontrolled studies have shown successful relief of migraine with metoclopramide of 75%. Further studies have reported success rate of 67% with IV metoclopramide. In this study the investigators seek to explore another option for treatment of headaches in the ED, one that may be more efficacious and efficient. Haloperidol (Haldol), a butyrophenone class of medication, is thought to act by affecting the dopamine 2 receptor in the brain. These receptors are relatively abundant in the brainstem nuclei and sympathetic ganglia and nerves, through which they may regulate autonomic visceral, gastrointestinal, and hemodynamic responses frequently associated with migraine. One study, demonstrated that 4 out of 5 patients felt significant relief in pain intensity with the use of haloperidol, even when other medications had failed. Relapses were rare, and several patients reported that haloperidol interrupted the prolonged, intractable migraine spiral they had suffered for days. Furthermore, a case series of six cases of migraine treated with 5mg of haloperidol IV after a 500 to 1000ml bolus of IV fluids reported complete or substantial relief within 25 to 65 minutes and side effects were reported as minimal.

The investigators hypothesize that Haloperidol is more efficacious than metoclopramide in the treatment of an acute headache or migraine in the ED in regard to a self-reported pain rating scale (Numeric Pain Intensity Scale), need for additional medication, emergency department return rates, and resolution of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present with a headache or migraine with onset less than or equal to 72 hours

Exclusion Criteria:

* Known pregnancy
* Breast-feeding women
* Known history of arrhythmias or QT prolongation (450 ms)
* Known adverse effects to haloperidol, diphenhydramine (Benadryl) or metoclopramide
* Subarachnoid hemorrhage
* Headaches caused by trauma, meningitis
* Congestive heart failure
* Parkinson's Disease
* Dementia
* Pheochromocytoma
* History of glaucoma
* History of seizures
* Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-02; Primary Completion 2017-04-24 (Actual); Study Completion 2017-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Lloyd, D.O., Principal Investigator — Attending Physician
Locations (1):
- OhioHealth Doctors Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metoclopramide (Reglan) | Haloperidol (Haldol)
Started | 35 | 31
Completed | 31 | 29
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metoclopramide (Reglan) | Haloperidol (Haldol) | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (9.9) | 36.9 (10.0) | 35.7 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Study was terminated early. Some baseline information entered for n=49 participants. Data not collected for 11 participants.
  Participants
    number analyzed (Participants) | 26 | 23 | 49
    Female | 8 | 9 | 17
    Male | 18 | 14 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Study was terminated early. Some baseline information entered for n=49 participants. Data not collected for 11 participants.
  Participants
    Race/Ethnicity: number analyzed (Participants) | 26 | 23 | 49
    Race/Ethnicity: Caucasian | 18 | 19 | 37
    Race/Ethnicity: African American | 6 | 4 | 10
    Race/Ethnicity: Somali | 1 | 0 | 1
    Race/Ethnicity: Hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60
Baseline Pain Score [Mean (Standard Deviation); unit: units on a scale] — Baseline Pain Score derived from Numeric Pain Intensity Scale. This scale is a patient-reported numeric measure of pain, from 0 [no pain] to 10 [worst pain imaginable.] Population: Study was terminated early. Some baseline information entered for n=49 participants. Data not collected for 11 participants.
  units on a scale
    number analyzed (Participants) | 26 | 23 | 49
    (all) | 8.13 (1.36) | 8.54 (1.34) | 8.35 (1.38)

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score According to the Numeric Pain Intensity Scale
Description: Numeric Pain Intensity scale is a standard rating tool for pain, ranging from 0-10, with 0=no pain and 10=worst pain imaginable.
Time Frame: Change from baseline (prior to treatment) to 1 hour post treatment (1 hour)
Population: Study was terminated early. Information entered for n=49 participants. Data not collected for 11 participants.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Metoclopramide (Reglan) | Haloperidol (Haldol)
Number analyzed (Participants) | 26 | 23
units on a scale | -2.86 (2.37) | -5.13 (2.59)

2. Secondary Outcome: Need for Additional Medications Used in the Emergency Department (ED)
Description: Need for additional medications in the ED will be evaluated via chart review at 48 hours post discharge
Time Frame: 48 hours post discharge
Population: Study was terminated early. Information entered for n=49 participants. Data not collected for 11 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Metoclopramide (Reglan) | Haloperidol (Haldol)
Number analyzed (Participants) | 26 | 23
Participants
  Yes | 7 | 4
  No | 4 | 9
  Unknown | 15 | 10

3. Secondary Outcome: Occurrence of Patient Return to the Emergency Department (ED) or Other Healthcare Provider for Headache/Migraine Within 48 Hours of ED Discharge
Description: Occurrence of patient return to the ED or other healthcare provider for headache/migraine within 48 hours of ED discharge will be evaluated via chart review at 48 hours post discharge
Time Frame: 48 hours post discharge
Population: Study was terminated early. Information entered for n=49 participants. Data not collected for 11 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Metoclopramide (Reglan) | Haloperidol (Haldol)
Number analyzed (Participants) | 26 | 23
Participants
  Yes | 0 | 0
  No | 26 | 23

ADVERSE EVENTS:
Time Frame: 48 hours
Description: Study was terminated early. Some information entered for n=49 participants. Data not collected for 11 participants.
Arm/Group | Metoclopramide (Reglan) | Haloperidol (Haldol)
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/23
Other Adverse Events (participants affected / at risk) | 0/26 | 0/23

LIMITATIONS AND CAVEATS:
This study was terminated by the IRB due to PI lapse in required training. Outcomes data reported includes preliminary figures for n=49 patients. Data not collected from 11 patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT02972502/Prot_SAP_000.pdf